CLINICAL TRIAL: NCT01038908
Title: Axillary Reverse Mapping in Breast Cancer
Brief Title: Breast Lymph Node Mapping
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: H09-00926
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node biopsy (SLNB); axillary lymph node dissection (ALND); lymphatics; blue dye
MeSH Terms: conditions — Breast Neoplasms | interventions — iso-sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Each patient will receive an injection of technetium-99m sulfur colloid directed subareolar or around the tumor. The material will be prepared as per manufacturer's specifications. The dose will be 20mBq given the same day of 80mBq given the day before. The Nuclear Medicine Department at St Paul's Hospital will perform the injection as per normal sentinel lymph node mapping protocol.
  Interventions: Other: Isosulfan Blue (Patent Blue Dye V)
- 2 (Active Comparator): Each patient will receive an injection of technetium-99m sulfur colloid directed subareolar or around the tumor. The material will be prepared as per manufacturer's specifications. The dose will be 20mBq given the same day of 80mBq given the day before. The Nuclear Medicine Department at St Paul's Hospital will perform the injection as per normal sentinel lymph node mapping protocol.
  Interventions: Other: Isosulfan Blue (Patent Blue Dye V)

INTERVENTIONS:
Other: Isosulfan Blue (Patent Blue Dye V) — 1. Inject radioactive isotope and scan for sentinel node (SLN) using gamma probe
  2. Pre-incision: SLN is identified
  3. Inject blue dye into patient's arm
  4. Complete procedure (SLNB and/or ALND)
  Arms: 1
Other: Isosulfan Blue (Patent Blue Dye V) — 1. Inject radioactive isotope and scan for sentinel node (SLN) using gamma probe
  2. Pre-incision: SLN is not identified (No localization)
  3. Inject blue dye into breast (nothing in arm)
  i. No localization: Inject blue dye into arm and perform ALND ii. Localization: Complete procedure (SLNB and/or ALND)
  Arms: 2

SUMMARY:
The purpose of this study is to map the arm lymphatic drainage system in the axilla with blue dye and the breast drainage system with a radioactive material. By identifying the arm lymphatics they can be protected during surgery and this may decrease the occurrence of lymphedema. The information obtained in this study may provide us with better surgical techniques to identify and protect the arm lymphatic drainage system in the axilla.

DETAILED DESCRIPTION:
This study is a non-randomized Phase II study of the Axillary Reverse Mapping (ARM) procedure for patients presenting with breast cancer requiring lymph node evaluation. The study will enroll 100 subjects, and will have two study arms: one for patients requiring only the SLNB procedure (roughly 67% of enrollees), and one for patients requiring a full ALND (roughly 33% of enrollees). For the analysis of study efficacy, each arm will be compared to its procedure-appropriate historical control for evidence of decrease in the 1-year lymphedema rate among patients undergoing SLNB or ALND.

Additional data will be collected on the treatment population's (a) variability in location of arm lymphatics, and (b) incidence of SLN crossover with arm lymphatics, along with success-rate data for identifying SLNs and arm lymphatics during SLNB and/or ALND. This additional data will add to our level of knowledge and experience regarding lymph node surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 19-100 years old
2. Not pregnant or breastfeeding
3. Breast cancer requiring LN evaluation for the breast
4. Willing participation following an informed consent process

Exclusion Criteria:

1. Patient < 19 y/o or > 100 y/o
2. Pregnant or breastfeeding
3. Allergy to blue dye
4. Locally advanced axillary disease
5. History of receiving neoadjuvant chemotherapy treatment
6. Prior axillary surgery or radiation therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Map arm lymphatic drainage system in the axilla | 4 years

SECONDARY OUTCOMES:
Decrease the occurrence of lymphedema | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Sam Wiseman, MD, FRCSC, FACS, Principal Investigator — University of British Columbia; Urve Kuusk, MD, FRCSC, Study Director — University of British Columbia; Carolyne Dingee, MD,FRCSC, Study Director — University of British Columbia; Elaine McKevitt, MD, FRCSC, Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - Mount Saint Joseph's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia